CLINICAL TRIAL: NCT02549625
Title: Phase I Safety and Feasibility Study of Intracoronary Delivery of Autologous Bone Marrow Derived Mononuclear Cells for Systemic, Single Right Ventricular Failure Due to Congenital Heart Disease
Brief Title: Phase I Safety and Feasibility Study of Intracoronary Delivery of Autologous Bone Marrow Derived Mononuclear Cells
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Timothy J Nelson, MD, PhD (Other)
Collaborators: Mayo Clinic (Other)
Responsible Party: Sponsor-Investigator, Timothy J Nelson, MD, PhD, Program Director, ReGen Theranostics, Inc.
Organization: ReGen Theranostics, Inc. (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-006427
Record Dates: First submitted 2015-09-10; First posted 2015-09-15 (Estimated); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Congenital Heart Disease
Keywords: Single right ventricular failure
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single-arm (Experimental): Intracoronary delivery of autologous bone marrow-derived mononuclear cells using catheterization procedure
  Interventions: Biological: Autologous Bone Marrow-derived Mononuclear Cells

INTERVENTIONS:
Biological: Autologous Bone Marrow-derived Mononuclear Cells
  Other Names: MNC

SUMMARY:
The objective of this study is to determine the safety and feasibility of autologous mononuclear cells (MNC) collected from bone marrow (BM) and intracoronary delivery for individuals with declining performance of their single right ventricle systemic pumps. This procedure has the potential to foster a new strategy for congenital heart patients. This is an open-label study of autologous MNC derived from bone marrow with a 2-year follow-up to document 1) related serious adverse events and 2) monitor changes in cardiac structure and function.

DETAILED DESCRIPTION:
This study is an open label Phase I trial to determine the safety and feasibility of bone marrow-derived mononuclear cells delivered into the coronary circulation of subjects with Fontan circulation and right ventricular dysfunction. Subjects will be screened at outpatient clinic visits at Mayo Clinic and interested qualified subjects will be consented and offered participation in this trial. Once informed consent has been obtained; preoperative values will be established and a selection committee will review subjects within three days prior to planned procedure to confirm inclusion and exclusion criteria. This will require a non-study cardiologist to review the clinical case and confirm the baseline cardiac function with evidence of disease progression with right ventricle dysfunction. However, individuals with decreased cardiac function requiring inotropic support and immediate listing for cardiac transplantation will NOT be included such that the risk of this research procedure may not be acceptable. Following cell-based product delivery, subjects will be followed for 6-months according to a pre-determined schedule that includes imaging studies along with questionnaires, electrophysiology and laboratory studies. Subjects will be contacted for an additional 18-months for surveillance by phone.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with Fontan circulation with right ventricular dysfunction
* Ejection fraction equal to or less than 40% despite optimal outpatient medical management for at least 3 months
* Able to undergo bone marrow aspirate according to clinical consultation with hematology (INR must be maintained at or below 1.5)
* Able to undergo an MRI or CT examination

Exclusion Criteria:

* Individuals or parents of minors unwilling to consent to participation
* Individuals with severe chronic diseases, extra-cardiac syndromes, or cancer
* Females 10 years and older with positive pregnancy test or lack of effective birth control method
* Individuals currently requiring IV inotropes
* Individuals with bleeding disorders or history of thrombosis
* Individuals not eligible for MRI and have elevated serum creatinine level (eGFR less that 45 mL/min) and therefore cannot have a CT examination
* Individuals not eligible for MRI and have a prior significant reaction to intravenous contrast required for CT examination
* Individuals with the following conditions within 60 days prior to procedure:

  * Cardiogenic shock or extracorporeal circulation;
  * New arrhythmia that required medication for control;
  * Documented infection requiring treatment with antibiotics, and/or current infection being treated with antibiotics;
  * Cardiac condition requiring emergency procedure;
  * Cardiovascular surgery;
  * Seizures or history of significant neurological injury;
  * Multi-system organ failure including acute or chronic renal failure

Ages: 2 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2015-08; Primary Completion 2020-11 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
Number of related serious adverse events | 6 months post cell delivery

SECONDARY OUTCOMES:
Number of subjects who died | 6 months post cell delivery
Number of subjects with sustained or symptomatic ventricular arrhythmias | 6 months post cell delivery
Number of subjects with acute decompensated heart failure | 6 months post cell delivery
Number of subjects with myocardial infarction | 6 months post cell delivery
Number of subjects with cardiac infection | 6 months post cell delivery
Number of subjects with unexpected cardiovascular procedures within 6 months following cellular transplantation | 6 months post cell delivery
Percentage of subjects that have cells delivered | 6 months post cell delivery
Percentage of subjects completing the 6-month follow-up | 6 months post cell delivery
Change in CT/MRI derived right ventricle ejection fraction | Baseline, 6 months post cell delivery
Change in diastolic ventricular volume | Baseline, 6 months post cell delivery
Change in systolic ventricular volume | Baseline, 6 months post cell delivery
Change in echocardiography derived right ventricle ejection fraction | Baseline, 6 months post cell delivery

CONTACTS AND LOCATIONS:
Overall Officials: Timothy J Nelson, M.D., Ph.D., Study Director — Mayo Clinic; Muhammad Y Qureshi, MBBS, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials